CLINICAL TRIAL: NCT05856032
Title: Effects of Using Acapella in Combination With Conventional Chest Physiotherapy Techniques to Improve Pulmonary Functions in Post CABG Patients.
Brief Title: Effects of Acapella With Conventional Chest Physiotherapy Techniques in Post CABG Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/MS-PT/01494
Record Dates: First submitted 2023-05-04; First posted 2023-05-12 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Cardiac Procedure Complication

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be blinded as they won't be knowing in which intervention group they are allocated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Use of Acapella device (Experimental): * Experimental group will receive treatment with Acapella device twice a day for 6 days post-operatively.
  * Participants in this group will also receive conventional chest physiotherapy protocol as: incentive spirometry, Active Cycles of Breathing Technique (ACBT), Diaphragmatic breathing exercises except manual chest physiotherapy techniques.
  Interventions: Device: Acapella device
- Conventional treatment (Active Comparator): •Participants in control or comparative group will receive conventional chest physiotherapy protocol as incentive spirometry, ACBT's, Diaphragmatic breathing exercises along with manual chest physiotherapy techniques as percussion and vibration.
  Interventions: Other: Conventional Treatment

INTERVENTIONS:
Device: Acapella device — Acapella is one of the Oscillatory Positive Expiratory Pressure (OPEP) device used in mobilization of peripheral secretions to the central trachea. It consists of a mouth piece and metal strip that is attached to a magnet which oscillates upon exhalation of the patient into the device results in oscillations. This helps in generating positive expiratory pressure (PEP) and oscillations of the magnetic ball assist in mucus collection and expectoration. Pulmonary functions are greatly reduced in patients undergone CABG surgery due to prolong effects of anaesthesia and muscle relaxants administered prior to surgery.
  Arms: Use of Acapella device
Other: Conventional Treatment — Conventional chest physiotherapy techniques
  Arms: Conventional treatment

SUMMARY:
To determine the effects of using Acapella as an oscillatory positive expiratory pressure device in combination with conventional chest physiotherapy for secretion removal and revival of pulmonary functions in hospitalized post coronary artery bypass grafting patients.

DETAILED DESCRIPTION:
Acapella is one of the Oscillatory Positive Expiratory Pressure (OPEP) device used in mobilization of peripheral secretions to the central trachea. It consists of a mouth piece and metal strip that is attached to a magnet which oscillates upon exhalation of the patient into the device results in oscillations. This helps in generating positive expiratory pressure (PEP) and oscillations of the magnetic ball assist in mucus collection and expectoration. Pulmonary functions are greatly reduced in patients undergone CABG surgery due to prolong effects of anesthesia and muscle relaxants administered prior to surgery. Ciliary motion along the pathway of pulmonary tract is depressed which results in decrease expectoration capacity, causes mucus retention and reduces pulmonary volumes and capacities. Chest physiotherapy is the treatment option for such patients that is being practiced over years. In recent years certain respiratory aids or devices are also in use to relieve secretion retention along with standard chest physiotherapy techniques.

The purpose of this study is to find the effects of using Acapella as an OPEP device along with conventional chest physiotherapy techniques in post-CABG surgery patients to relieve mucus retention and improving pulmonary functions post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders within age range of 45-65 years
* Elective CABG surgery patients
* Patients undergoing Phase 1 cardiac rehabilitation post CABG
* Patients who are vitally stable post operatively

Exclusion Criteria:

* Patient having prolong intubation period post-operatively
* Patients having long term arrythmias prior to surgery
* Patients having an implanted pacemaker
* Patients having uncontrolled diabetes, sepsis or any metabolic condition
* Patients with impaired cognition.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Change in Forced Expiratory Volume in 1 second | pre-operative day 1 and post-operative day 6 of CABG surgery
  Forced expiratory volume in 1 second, measures the volume of air that is expired into the mouthpiece of the digital spirometer in first second after full inhalation. Normally ranges between 80% to 120% of average predicted values
Change in Forced Vital Capacity | pre-operative day 1 and post-operative day 6 of CABG surgery
  FVC: forced vital capacity, measures the volume of air blown forcefully into the mouthpiece following full inhalation. Normal values ranges between 80% to 120% of average predicted values
Ratio of Forced Expiratory Volume in 1 second and Forced Vital Capacity | pre-operative day 1 and post-operative day 6 of CABG surgery
  FEV1/FVC: the FEV1/FVC ratio is calculated by dividing measured FEV1 value by measured FVC value. In a healthy individual it ranges between 70 to 85%.

SECONDARY OUTCOMES:
Borg dyspnoea scale | 6th post-operative day after CABG surgery
  A scale used to measure level of exhaustion, breathlessness and fatigue during physical work. Patients are asked to rate the level of physical exertion, fatigue and dyspnoea on a 6-20 scale where 6 shows no fatigue at all and 20 indicates maximum exertion and fatigue.
Amount of secretions expectorated | 6th post-operative day after CABG surgery
  tracing the amount of pulmonary secretions produced per day as a result of using respiratory aids along with conventional chest physiotherapy techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Malik Muhammad Ali Awan, MSPT, Principal Investigator — Riphah International University
Locations (1):
- Armed Forces Institute of Cardiology, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No